CLINICAL TRIAL: NCT01889862
Title: A Four-Part, Phase 3, Randomized, Double-Blind, Placebo- Controlled, Four-Arm, Discontinuation Study to Evaluate the Efficacy and Safety of Subcutaneous Injections of BMN 165 Self-Administered by Adults With Phenylketonuria (PKU)
Brief Title: Phase 3 Study to Evaluate the Efficacy & Safety of Self-Administered Injections of BMN165 by Adults With PKU
Acronym: Prism-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 165-302
Record Dates: First submitted 2013-06-18; First posted 2013-07-01 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU; PEG-PAL; Prism; BioMarin; rAvPAL-PEG; BMN165
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase; Dextrans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BMN165 20mg/day (Active Comparator): BMN165 20mg/day self-administered daily
  Interventions: Drug: BMN165 20mg/day
- 20 mg/day Placebo (Placebo Comparator): 20 mg/day Placebo self-administered daily
  Interventions: Drug: Placebo
- BMN165 40mg/day (Active Comparator): BMN165 40mg/day self-administered daily
  Interventions: Drug: BMN165 40mg/day
- 40 mg/day Placebo (Placebo Comparator): 40 mg/day Placebo self-administered daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMN165 20mg/day — BMN165 20mg/day self-administered daily
  Other Names: PEG-PAL
  Arms: BMN165 20mg/day
Drug: BMN165 40mg/day — BMN165 40mg/day self-administered daily
  Other Names: PEG-PAL
  Arms: BMN165 40mg/day
Drug: Placebo — Non-drug placebo, self-administered daily
  Other Names: Dextran 40
  Arms: 20 mg/day Placebo; 40 mg/day Placebo

SUMMARY:
The BMN 165 clinical development program has been designed to demonstrate the safety and efficacy of BMN 165 in reducing blood Phe concentrations in adults with PKU.

DETAILED DESCRIPTION:
165-302 is a Phase 3, 4 Part, Randomized, Double-Blind, Placebo-Controlled, Discontinuation Study to Evaluate the Efficacy and Safety of Self Administered Subcutaneous Injections of BMN 165 by Adults With PKU.

This study is open only to adults who have been exposed to BMN165 in a previous study.

Study BMN 165-302 is a four-Part, Phase 3 study.

* Part 1: Open-label period
* Part 2: A Randomized, double-blind, placebo-controlled period of 8 weeks
* Part 3: Two sub-Parts to Part 3:- Part 3A - BMN 165 administered using vial and syringe during this open label period. Part 3B - BMN 165 administered using prefilled syringe during this open-label period.
* Part 4: A long-term, open-label extension period.

ELIGIBILITY:
INCLUSION CRITERIA

Individuals eligible to participate in this study must meet all of the following criteria:

* Have completed a prior BMN 165 study (PAL-003, 165-205, or 165-301) prior to screening
* Have had a stable BMN 165 dose regimen for at least 14 days prior to screening
* Are at least 18 y/o and no older than 70 y/o at screening

  * Subjects who are < 18 y/o and are already enrolled into Study 165-301 under Amendment #1 (10JAN2014) may enroll into this study
* Has identified a person who is > 18 y/o who has the neurocognitive and linguistic capacities to comprehend and complete the Profile of Mood States (POMS)-Observer rated scale
* Has identified a competent person(s) > 18 y/o who can observe the subject during study drug administration at certain points in the study

  * A home healthcare nurse may perform the study drug observations
* Are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures; for minors, parent or guardian provides written consent and assent may be requested
* Are willing and able to comply with all study procedures
* For females of childbearing potential, a negative pregnancy test at screening and willing to have additional pregnancy tests during the study
* If sexually active, willing to use two acceptable methods of contraception during and for 4 weeks after the study

  * Males post vasectomy for 2 years with no known pregnancies do not need to use any other forms of contraception during the study.
  * Females who have been in menopause for at least 2 years, have had a tubal ligation at least 1 year prior to screening, or have had a total hysterectomy do not need to use any other forms of contraception during the study.
* Have received documented approval from a study dietitian confirming that the subject is capable of maintaining their diet
* Have neurocognitive and linguistic capacities to comprehend and answer investigator's prompts for the Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) Investigator rated instrument and to complete the POMS-Subject rated scale
* If applicable, maintained stable dose of medication for Attention Deficit Hyperactivity Disorder (ADHD), depression, anxiety, or other psychiatric disorder ≥8 weeks prior to enrollment and willing to maintain stable dose throughout study unless a change is medically indicated
* General good health, as evidenced by physical examination, clinical laboratory evaluations, and ECG tests at screening

Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

* Use of any investigational product (except BMN 165) or investigational medical device within 30 days prior to screening or requirement for any investigational agent prior to completion of all scheduled study assessments
* Use of any medication (except BMN 165) intended to treat PKU, including the use of large neutral amino acids, within 2 days prior to the administration of study drug
* Have known hypersensitivity to Dextran® or components of Dextran
* Use or planned use of any injectable drugs containing PEG (except for BMN 165), including medroxyprogesterone injection, within 3 months prior to screening and during study participation
* Current use of levodopa
* A positive test for HIV antibody, hepatitis B surface antigen, or hepatitis C antibody
* A history of organ transplantation or taking chronic immunosuppressive therapy
* A history of substance abuse in the past 12 months or current alcohol or drug abuse
* Current participation in the Kuvan registry study (PKUDOS). Patients may discontinue the PKUDOS registry trial to allow enrollment in this study
* Pregnant or breastfeeding at screening or planning to become pregnant (self or partner) or breastfeed at any time during the study
* Concurrent disease or condition that would interfere with study participation or safety.
* Major surgery planned during the study period
* Any condition that in the view of the investigator, places the subject at high risk of poor treatment compliance or terminating early from the study
* Alanine aminotransferase (ALT) concentration at least 2x the upper limit of normal
* Creatinine at least 1.5x the upper limit of normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2016-01-13 (Actual); Study Completion 2019-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Specialist, Study Director — BioMarin Pharmaceutical
Locations (29):
- United States (29):
  - University of California, San Diego Clinical and Translational Research Institute, La Jolla, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida Clinical Research Center, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory Universty, Department of Human Genetics, Division of Medical Genetics, Atlanta, Georgia
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - Wayne State University Clinical Research Center at the Mott Center, Detroit, Michigan
  - University of Missouri Health Center, Columbia, Missouri
  - Washington University Center for Applied Research Sciences, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper Health Systems, Camden, New Jersey
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - Icahn School of Medicine at Mount Sinai Medical Center, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas Houston Medical School, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Washinton, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilder DA, Arnold GL, Dimmock D, Grant ML, Janzen D, Longo N, Nguyen-Driver M, Jurecki E, Merilainen M, Amato G, Waisbren S. Improved attention linked to sustained phenylalanine reduction in adults with early-treated phenylketonuria. Am J Med Genet A. 2022 Mar;188(3):768-778. doi: 10.1002/ajmg.a.62574. Epub 2021 Nov 26. PMID 34826353
- See also: BioMarin sponsored PKU educational/community website — http://www.pku.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study, conducted in 29 study centers of United States.
Pre-assignment Details: A total of 51 out of 215 subjects entered Part 4 directly from 165-301, as they did not receive target dose of 20 or 40 mg/day in 165-301.
Groups:
- BMN165 20mg/Day: BMN165 20mg/day subcutaneous injection administered using vial and syringe in Part 1, 2 and 3A.
  BMN165 20mg/day subcutaneous injection administered using a prefilled syringe in Part 3B.
- Placebo 20mg/Day: Matching placebo 20mg/day subcutaneous injection administered using vial and syringe in Part 2.
- BMN165 40mg/Day: BMN165 40mg/day subcutaneous injection administered using vial and syringe in Part 1, 2 and 3A.
  BMN165 40mg/day subcutaneous injection administered using a prefilled syringe in Part 3B.
- Placebo 40mg/Day: Matching placebo 40mg/day subcutaneous injection administered using vial and syringe in Part 2.
- BMN165: Up to 60mg/day BMN165 subcutaneous injection administered using a prefilled syringe in Part 4.
Period: Part 1 (Up to 13 Weeks)
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day | BMN165
Started (51 subjects out of 215 entered Part 4 directly, as they didn't receive target dose in study 165-301.) | 86 | 0 | 78 | 0 | 0
Completed (57 Subjects out of 164 didn't meet Part 2 eligibility criterion, so transitioned directly to Part 4) | 74 (Out of 164, total 12 subjects have not completed Part 1.) | 0 | 78 | 0 | 0
Not Completed | 12 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Period: Part 2 (8 Weeks)
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day | BMN165
Started | 34 (Subjects ≥20% reduction in blood Phe from naïve baseline levels are randomized in Part 2.) | 15 (Subjects ≥20% reduction in blood Phe from naïve baseline levels are randomized in Part 2.) | 32 (Subjects ≥20% reduction in blood Phe from naïve baseline levels are randomized in Part 2.) | 14 (Subjects ≥20% reduction in blood Phe from naïve baseline levels are randomized in Part 2.) | 0
Per Amendment #2 of the Protocol (Subjects not included in mITT, if the last two consecutive blood Phe reduction of ≥ 20% in Part 1.) | 29 | 14 | 29 | 14 | 0
Completed (5 subjects unable to complete Part 2 due to an Adverse Event transitioned directly into Part 4.) | 34 | 15 | 31 | 14 | 0
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: Part 3A/B (6 Week)
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day | BMN165
Started | 48 (Subjects switch from placebo to active 20mg/kg.) | 0 (Subjects switch from placebo to active 20mg/kg.) | 41 (Subjects switch from placebo to active 40mg/kg.) | 0 (Subjects switch from placebo to active 40mg/kg.) | 0
Per Amendment #2 of the Protocol (58 of 89 subjects enrolled under Amendment #2 were included in the PK/PD analyses.) | 34 | 0 | 26 | 0 | 0
Completed | 48 | 0 | 41 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 4 (Up to 274 Weeks)
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day | BMN165
Started | 0 (51, 57, 5 and 89 subjects from 165-301, 165-302 Part 1, 2 & 3 entered 165-302 Part 4 respectively.) | 0 | 0 (51, 57, 5 and 89 subjects from 165-301, 165-302 Part 1, 2 & 3 entered 165-302 Part 4 respectively.) | 0 | 202 (Total of 202 subjects from 165-301, Part 1, 2, 3 entered Part 4 to receive dose of up to 60mg/kg.)
Completed | 0 | 0 | 0 | 0 | 172
Not Completed | 0 | 0 | 0 | 0 | 30
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 5
Not completed — Subject withdrew consent | 0 | 0 | 0 | 0 | 14
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 5
Not completed — Protocol deviations | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All Subjects consists of subjects participated in 165-302 Part 1, 2, 3 and 4.
Groups:
- All Subjects: BMN165 20mg/Day:
  BMN165 20mg/day subcutaneous injection administered using vial and syringe in Part 1, 2 and 3A.
  BMN165 20mg/day subcutaneous injection administered using a prefilled syringe in Part 3B.
  Placebo 20mg/Day:
  Matching placebo 20mg/day subcutaneous injection administered using vial and syringe in Part 2.
  BMN165 40mg/Day:
  BMN165 40mg/day subcutaneous injection administered using vial and syringe in Part 1, 2 and 3A.
  BMN165 40mg/day subcutaneous injection administered using a prefilled syringe in Part 3B.
  Placebo 40mg/Day:
  Matching placebo 40mg/day subcutaneous injection administered using vial and syringe in Part 2.
  BMN165:
  Up to 60mg/day BMN165 subcutaneous injection administered using a prefilled syringe in Part 4.
Arm/Group | All Subjects
Number analyzed (Participants) | 215
Age, Continuous [Mean (Standard Deviation); unit: yrs] | 29.22 (8.74)
Age, Customized [Count of Participants; unit: Participants]
  16 - <18 years | 11
  18 - <66 years | 204
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  White | 211
  Black/African American | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Blood Plasma Phenylalanine (Phe) Concentration at Part 2
Description: Blood phe concentration in subjects previously exposed to BMN165 who were administered BMN165 20 or 40 mg/day compared with those who were administered a matching placebo.
Time Frame: At Part 2 baseline and change from baseline at Part 2 week 8
Population: Modified Intent-to-Treat (mITT) population consists of all subjects who reached the randomized dose of 20mg/day or 40mg/day and were randomized into Part 2 with a mean blood Phe reduction of ≥20% (using the last two consecutive blood Phe assessments of Part 1) from the baseline of 165-301 (or the Phase 2 study in which they initiated BMN165).
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day
Number analyzed (Participants) | 29 | 14 | 29 | 14
µmol/L
  Part 2 Baseline | 596.8 (582.75) | 563.9 (504.62) | 410.9 (439.95) | 508.2 (363.68)
  Change from Baseline Part 2 Week 8 | -65.9 (192.02) | 996.4 (555.00) | 114.1 (332.40) | 599.0 (507.40)
Statistical Analysis 1: Comparison: BMN165 20mg/Day vs Placebo 20mg/Day; Change in blood Phe concentration during Part 2 in subjects previously exposed to BMN165 who self administer BMN165 20mg/day compared with those who self administer matching placebo; Test type: Superiority; p < 0.0001, ANCOVA — Based on Mixed-Effect Model Repeated Measure (MMRM) model with change from baseline as the response variable, and treatment, visit and treatment by visit interaction and baseline blood phe concentration as factors; Mean Difference (Net) = -973.02, 95% CI 2-sided [-1204.19 to -741.85]
Statistical Analysis 2: Comparison: BMN165 40mg/Day vs Placebo 40mg/Day; Change in blood Phe concentration during Part 2 in subjects previously exposed to BMN165 who self administer BMN165 40mg/day compared with those who self administer matching placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -588.50, 95% CI 2-sided [-830.07 to -346.94]

2. Secondary Outcome: Change From Baseline in the Cognitive and Mood Symptoms Measured by ADHD Rating Scale (RS)-IV Inattention Subscale at Part 2
Description: Attention deficit hyperactivity disorder rating scale IV (ADHD RS-IV) is investigator-rated, 9-item, inattention subscale score ranges from 0 to 27, with higher scores indicative of a greater degree of impairment and a baseline score >9 indicative of a presence of symptoms.
Time Frame: At Part 2 baseline and change from baseline at Part 2 week 8
Population: mITT population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day
Number analyzed (Participants) | 29 | 14 | 29 | 14
Units on a scale
  Baseline | 5.9 (4.70) | 5.0 (4.26) | 6.0 (6.45) | 2.9 (3.68)
  Change from Baseline Part 2 Week 8 | 1.1 (3.96) | 1.2 (3.00) | 0.5 (5.36) | -0.4 (3.44)

3. Secondary Outcome: Change From Baseline in the Blood Plasma Phenylalanine (Phe) Concentration at Part 4
Description: The long term effect of multiple dose levels of BMN165 on blood phe concentration in subjects who are administered BMN165 using pre-filled syringes.
Time Frame: At Part 4 week 57, 105, 161, 209 and 249
Population: All Subjects Entered 165-302 Part 4 Data
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- BMN165 < 20 mg/Day - Part 4; BMN165 20 to < 40 mg/Day - Part 4: BMN165 < 20 mg/day subcutaneous injection administered using a prefilled syringe in Part 4.
- BMN165 40 to < 60 mg/Day - Part 4: BMN165 40 to < 60 mg/day subcutaneous injection administered using a prefilled syringe in Part 4.
- BMN165 >= 60 mg/Day - Part 4: BMN165 >= 60 mg/day subcutaneous injection administered using a prefilled syringe in Part 4.
- BMN165 All Dose - Part 4: Up to 60mg/day BMN165 subcutaneous injection administered using a prefilled syringe in Part 4.
Arm/Group | BMN165 < 20 mg/Day - Part 4 | BMN165 20 to < 40 mg/Day - Part 4 | BMN165 40 to < 60 mg/Day - Part 4 | BMN165 >= 60 mg/Day - Part 4 | BMN165 All Dose - Part 4
Number analyzed (Participants) | 61 | 131 | 184 | 62 | 202
µmol/L
  Change from Baseline to Part 4 Week 57: number analyzed (Participants) | 20 | 36 | 91 | 33 | 180
  Change from Baseline to Part 4 Week 57 | -1004.9 (541.19) | -984.0 (531.33) | -810.2 (595.24) | -662.3 (465.61) | -839.5 (562.74)
  Change from Baseline to Part 4 Week 105: number analyzed (Participants) | 29 | 31 | 74 | 32 | 166
  Change from Baseline to Part 4 Week 105 | -1015.3 (557.00) | -1109.2 (474.25) | -858.5 (593.73) | -641.0 (568.67) | -890.8 (578.38)
  Change from Baseline to Part 4 Week 161: number analyzed (Participants) | 14 | 29 | 31 | 22 | 96
  Change from Baseline to Part 4 Week 161 | -1006.5 (514.76) | -1111.9 (519.40) | -662.8 (433.80) | -808.6 (558.22) | -882.0 (528.61)
  Change from Baseline to Part 4 Week 209: number analyzed (Participants) | 8 | 5 | 8 | 9 | 30
  Change from Baseline to Part 4 Week 209 | -897.3 (494.41) | -1020.4 (495.79) | -541.6 (245.83) | -961.7 (339.92) | -842.3 (418.37)
  Change from Baseline to Part 4 Week 249: number analyzed (Participants) | 2 | 0 | 0 | 1 | 3
  Change from Baseline to Part 4 Week 249 | -1059.5 (160.51) |  |  | -1314.0 (NA) — Number of subjects participated in week 249 visit is one. | -1144.3 (185.67)

4. Secondary Outcome: Change From Baseline in the Cognitive and Mood Symptoms Measured by PKU POMS TMD at Part 2
Description: Phenylketonuria (PKU) Total Mood Disturbance (TMD) Profile of Mood States (POMS)
  PKU POMS TMD is self-rated, each item in the tool is rated using a five-point Likert scale: 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a bit), and 4 (extremely).
Time Frame: At Part 2 baseline and change from baseline at Part 2 week 8
Population: mITT population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day
Number analyzed (Participants) | 29 | 14 | 29 | 14
Units on a scale
  Baseline | 7.1 (14.18) | 8.6 (10.84) | 8.9 (12.28) | 5.0 (8.56)
  Change from Baseline Part 2 Week 8 | 4.8 (12.63) | 4.3 (11.96) | -2.0 (10.25) | 0.0 (14.08)

5. Secondary Outcome: Change From Baseline in the Cognitive and Mood Symptoms Measured by PKU POMS Confusion Subscale at Part 2
Description: PKU POMS confusion mood domain (referred to as the confusion subscale) is self-rated, each item in the tool is rated using a five-point Likert scale: 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a bit), and 4 (extremely).
Time Frame: At Part 2 baseline and change from baseline at Part 2 week 8
Population: mITT population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day
Number analyzed (Participants) | 29 | 14 | 29 | 14
Units on a scale
  Baseline | 2.0 (2.09) | 2.1 (1.49) | 2.4 (2.02) | 1.2 (1.53)
  Change from Baseline Part 2 Week 8 | 0.8 (2.79) | 1.4 (2.47) | -0.3 (1.84) | 0.5 (2.22)

6. Secondary Outcome: Change From Baseline in the Cognitive and Mood Symptoms Measured by POMS TMD at Part 2
Description: Full-length POMS TMD is self-rated, each item in the tool is rated using a five-point Likert scale: 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a bit), and 4 (extremely).
Time Frame: At Part 2 baseline and change from baseline at Part 2 week 8
Population: mITT population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | BMN165 20mg/Day | Placebo 20mg/Day | BMN165 40mg/Day | Placebo 40mg/Day
Number analyzed (Participants) | 29 | 14 | 29 | 14
Units on a scale
  Baseline | 16.2 (35.63) | 18.1 (28.26) | 24.3 (35.38) | 13.3 (21.63)
  Change from Baseline Part 2 Week 8 | 13.1 (30.73) | 7.3 (26.23) | -3.2 (26.63) | -1.7 (29.34)

ADVERSE EVENTS:
Time Frame: Up to 301 weeks
Description: Safety Analyses consists of the population for safety analyses of all subjects who enrolled into the study and all subjects who enrolled into each study part for analysis by study part.
Groups:
- Part 1 - 20 mg/Day; Part 2 - 20 mg/Day Active: BMN165 20mg/day subcutaneous injection administered using vial and syringe.
- Part 1 - 40 mg/Day; Part 2 - 40 mg/Day Active: BMN165 40mg/day subcutaneous injection administered using vial and syringe.
- Part 2 - 20 mg/Day Placebo: Matching placebo 20mg/day subcutaneous injection administered using vial and syringe.
- Part 2 - 40 mg/Day Placebo: Matching placebo 40mg/day subcutaneous injection administered using vial and syringe.
- Part 3 - Stay on Active 20 mg/Day; Part 3 - Switch From Placebo to Active 20 mg/Day: BMN165 20mg/day subcutaneous injection administered using vial and syringe in Part 3A.
  BMN165 20mg/day subcutaneous injection administered using a prefilled syringe in Part 3B.
- Part 3 - Stay on Active 40 mg/Day; Part 3 - Switch From Placebo to Active 40 mg/Day: BMN165 40mg/day subcutaneous injection administered using vial and syringe in Part 3A.
  BMN165 40mg/day subcutaneous injection administered using a prefilled syringe in Part 3B.
- Part 4 - < 20 mg/Day: BMN165 <20mg/day subcutaneous injection administered using a prefilled syringe.
- Part 4 - 20 to < 40 mg/Day: BMN165 20 to <40mg/day subcutaneous injection administered using a prefilled syringe.
- Part 4 - 40 to < 60 mg/Day: BMN165 40 to <60mg/day subcutaneous injection administered using a prefilled syringe.
- Part 4 - >= 60 mg/Day: BMN165 >=60mg/day subcutaneous injection administered using a prefilled syringe.
Arm/Group | Part 1 - 20 mg/Day | Part 1 - 40 mg/Day | Part 2 - 20 mg/Day Active | Part 2 - 40 mg/Day Active | Part 2 - 20 mg/Day Placebo | Part 2 - 40 mg/Day Placebo | Part 3 - Stay on Active 20 mg/Day | Part 3 - Stay on Active 40 mg/Day | Part 3 - Switch From Placebo to Active 20 mg/Day | Part 3 - Switch From Placebo to Active 40 mg/Day | Part 4 - < 20 mg/Day | Part 4 - 20 to < 40 mg/Day | Part 4 - 40 to < 60 mg/Day | Part 4 - >= 60 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/78 | 0/34 | 0/32 | 0/15 | 0/14 | 0/23 | 0/18 | 0/11 | 0/8 | 0/67 | 0/152 | 0/186 | 0/89
Serious Adverse Events (participants affected / at risk) | 6/86 | 2/78 | 0/34 | 2/32 | 1/15 | 0/14 | 1/23 | 0/18 | 0/11 | 0/8 | 7/67 | 6/152 | 16/186 | 5/89
Other Adverse Events (participants affected / at risk) | 70/86 | 59/78 | 27/34 | 28/32 | 14/15 | 13/14 | 19/23 | 15/18 | 8/11 | 7/8 | 62/67 | 105/152 | 178/186 | 59/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - 20 mg/Day (N=86) | Part 1 - 40 mg/Day (N=78) | Part 2 - 20 mg/Day Active (N=34) | Part 2 - 40 mg/Day Active (N=32) | Part 2 - 20 mg/Day Placebo (N=15) | Part 2 - 40 mg/Day Placebo (N=14) | Part 3 - Stay on Active 20 mg/Day (N=23) | Part 3 - Stay on Active 40 mg/Day (N=18) | Part 3 - Switch From Placebo to Active 20 mg/Day (N=11) | Part 3 - Switch From Placebo to Active 40 mg/Day (N=8) | Part 4 - < 20 mg/Day (N=67) | Part 4 - 20 to < 40 mg/Day (N=152) | Part 4 - 40 to < 60 mg/Day (N=186) | Part 4 - >= 60 mg/Day (N=89)
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Anaphylactoid Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brief Psychotic Disorder with Marked Stressors (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parasomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epiploic Appendagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoid Tissue Hyperplasia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendix Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Xanthogranuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - 20 mg/Day (N=86) | Part 1 - 40 mg/Day (N=78) | Part 2 - 20 mg/Day Active (N=34) | Part 2 - 40 mg/Day Active (N=32) | Part 2 - 20 mg/Day Placebo (N=15) | Part 2 - 40 mg/Day Placebo (N=14) | Part 3 - Stay on Active 20 mg/Day (N=23) | Part 3 - Stay on Active 40 mg/Day (N=18) | Part 3 - Switch From Placebo to Active 20 mg/Day (N=11) | Part 3 - Switch From Placebo to Active 40 mg/Day (N=8) | Part 4 - < 20 mg/Day (N=67) | Part 4 - 20 to < 40 mg/Day (N=152) | Part 4 - 40 to < 60 mg/Day (N=186) | Part 4 - >= 60 mg/Day (N=89)
Nasopharyngitis (Infections and infestations) | 7 | 11 | 4 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 15 | 27 | 59 | 19
Upper respiratory tract infection (Infections and infestations) | 8 | 5 | 1 | 0 | 3 | 2 | 3 | 2 | 1 | 0 | 14 | 29 | 51 | 10
Sinusitis (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 9 | 13 | 22 | 11
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 5 | 15 | 8
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 9 | 13 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 11 | 7
Urinary tract infection (Infections and infestations) | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 5 | 13 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 10 | 4
Ear infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 4 | 6 | 3
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 10 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 6 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 6 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 3
Injection site reaction (General disorders) | 13 | 7 | 4 | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 6 | 14 | 46 | 11
Injection site bruising (General disorders) | 9 | 7 | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 5 | 14 | 41 | 12
Injection site pruritus (General disorders) | 6 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 9 | 24 | 10
Fatigue (General disorders) | 8 | 3 | 4 | 3 | 3 | 0 | 5 | 4 | 0 | 1 | 10 | 8 | 14 | 10
Injection site induration (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 14 | 24 | 6
Injection site pain (General disorders) | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 22 | 9
Injection site swelling (General disorders) | 5 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 9 | 19 | 3
Injection site erythema (General disorders) | 4 | 5 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 19 | 7
Pyrexia (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 19 | 6
Peripheral swelling (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 15 | 2
Pain (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 2 | 10 | 5
Injection site mass (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 12 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 10 | 1
Injection site haemorrhage (General disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 5 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 13 | 7 | 2 | 1 | 2 | 3 | 0 | 3 | 2 | 16 | 33 | 64 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 10 | 14 | 33 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 9 | 14 | 24 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 16 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 5 | 15 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 12 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 5
Headache (Nervous system disorders) | 16 | 12 | 6 | 2 | 3 | 4 | 2 | 3 | 1 | 0 | 20 | 29 | 59 | 24
Dizziness (Nervous system disorders) | 2 | 7 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 10 | 6 | 21 | 11
Migraine (Nervous system disorders) | 3 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 6 | 8 | 18 | 9
Disturbance in attention (Nervous system disorders) | 0 | 0 | 4 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 5 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 8 | 1
Memory impairment (Nervous system disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 2 | 3 | 1 | 0 | 2 | 2 | 0 | 1 | 7 | 8 | 34 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7 | 1 | 4 | 0 | 1 | 1 | 1 | 1 | 0 | 6 | 13 | 33 | 14
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 12 | 28 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 5 | 12 | 12 | 6
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 9 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 8 | 4
Vomiting (Gastrointestinal disorders) | 4 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 8 | 18 | 34 | 13
Nausea (Gastrointestinal disorders) | 5 | 5 | 4 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 10 | 11 | 28 | 16
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 8 | 15 | 25 | 9
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 5 | 17 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 10 | 10 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 7 | 10 | 6
Toothache (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 6 | 12 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 6 | 8 | 9
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 10 | 6
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 11 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 6 | 20 | 29 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 14 | 32 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 9 | 12 | 20 | 8
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 5 | 12 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 7 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 3 | 1 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 9 | 9 | 22 | 5
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 12 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 7 | 5
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 8 | 2
Amino acid level decreased (Investigations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 9 | 13 | 37 | 13
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 6 | 1
Complement factor C3 decreased (Investigations) | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 5 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 4 | 3 | 0 | 2 | 1 | 1 | 1 | 0 | 11 | 10 | 23 | 6
Depression (Psychiatric disorders) | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 9 | 11 | 13 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 17 | 2
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 1
Seasonal allergy (Immune system disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 8 | 6 | 19 | 3
Hypersensitivity (Immune system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 10 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 5 | 1 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 4 | 9 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 5 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 8 | 18 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Depressive symptom (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Dyspraxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Distractibility (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperreflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 5 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood cortisol decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 6 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 6 | 0
Complement factor decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days